CLINICAL TRIAL: NCT05046587
Title: Characterization of Suicidal Depression Within a Large Cohort of Inpatients: a One-year Prospective Study.
Brief Title: Characterization of Suicidal Depression
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0395
Record Dates: First submitted 2021-07-05; First posted 2021-09-16 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Depression
Keywords: Suicide; Suicidal Ideation; Suicidal Depression
MeSH Terms: conditions — Depression; Suicide; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antidepressants are widely used to prevent suicidal risk. However, even though the use of antidepressants has been associated with a 40-60% decrease in suicidal risk, they do not seem to be sufficient and appropriate. Indeed recent studies have shown that patients with a history of suicide attempt and/or with current suicidal ideation (SI) respond less well to antidepressant treatments. This suggests that patients with depression with SI may be different from those with depression without SI, thus requiring specific treatments for both SI reduction and depressive remission. In other words, suicidal depression may be a specific subtype of depression.

The study aims to characterize the clinical phenotype of patients with suicidal depression vs. those without suicidal depression, and to assess the occurrence of suicidal events at one year in patients with suicidal depression vs. without suicidal depression.

All data having already been collected during the particpation of patients in various clinical research studies of the department

ELIGIBILITY:
Inclusion criteria:

* Over 18 years old
* Hospitalization in the Department of Emergency Psychiatry and Acute Care (Montpellier University Hospital) between 2012 and 2019
* Having being enrolled in one the department's clinical studies between 2012 and 2019
* Moderate to severe characterized depressive episode according to DSM-5 diagnostic criteria (severity assessed with BDI, IDSC-30 and QIDS)

Exclusion criteria:

* Protection by law (guardianship or curatorship)
* Deprivation of liberty (by judicial or administrative decision)
* Bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depressed patients with and without suicidal ideation, admitted to the Department of Emergency Psychiatry and Acute Care (Montpellier University Hospital) and enrolled in one of the department's clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 898 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
characterization of the patient clinical phenotype | day 1
  characterization of the patient clinical phenotype

SECONDARY OUTCOMES:
Suicidal events at one year | 1 year
  Occurrence of suicidal events (actual, interrupted and aborted or self-aborted suicide attempts) assessed with C-SSRS suicidal behaviour subscale (4 yes/no questions)
Hospitalization for suicidal ideation | 1 year
  Occurrence of hospitalization for suicidal ideation, based on the patient medical record
Suicidal events at one year | 1 year
  Occurrence of suicidal events (actual, interrupted and aborted or self-aborted suicide attempts) based on the patient medical records

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte NOBILE, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC